CLINICAL TRIAL: NCT03768544
Title: Generalized Anxiety Disorder in Older Adults : Efficacy of a Self-help Treatment Guided by Trained Lay Providers
Brief Title: Self-help Guided by Lay Providers for Anxiety in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); CIUSSS du Centre-Sud-de-l'Île-Montréal (Unknown); Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke (Other); Integrated University Health and Social Services Center of the Capitale-Nationale (Other)
Responsible Party: Principal Investigator, Philippe Landreville, Full professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIRUL 118715
Record Dates: First submitted 2018-11-21; First posted 2018-12-07 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Generalized Anxiety Disorder
Keywords: generalized anxiety disorder; older adult; psychological treatment; randomized controlled trial
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Treatment Delay

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-help guided by a lay provider (Experimental)
  Interventions: Behavioral: Self-help guided by a lay provider
- Waiting list where participants wait for delayed treatment (Other)
  Interventions: Behavioral: Self-help guided by a lay provider; Behavioral: Waiting list where participants wait for delayed treatment

INTERVENTIONS:
Behavioral: Self-help guided by a lay provider — Self-help based on the principles of cognitive-behavioral therapy and guided by a lay provider. Treatment lasts 15 weeks, is based on a participant's manual, and consists of relaxation, differentiation of the main types of worries, learning to tolerate uncertainty, questioning false beliefs about worries, problem solving, cognitive exposure, and planning pleasant activities. Weekly telephone sessions with the lay provider serve to provide support.
Behavioral: Waiting list where participants wait for delayed treatment — Participants have a 15-week wait period during which they receive a 15-minute telephone call from the local professional research assistant on three occasions separated by four-week intervals. The purpose of these calls is to encourage the participant to persevere until the start of treatment and to identify potential negative effects that could be associated with the waiting period. Participants receive self-help guided by a lay provider after the waiting period.
  Arms: Waiting list where participants wait for delayed treatment

SUMMARY:
Few older adults receive treatment for Generalized Anxiety Disorder (GAD) despite a high prevalence in this population and significant associated health care costs. Although older adults generally prefer psychotherapy to medication for help with anxiety, face-to-face psychotherapy is difficult to access for many of them. Psychological guided self-help (GSH), which patients use by themselves at home under the supervision of a licensed mental health provider (e.g., psychologist), has been shown to be effective. However, the capacity of our health care system to respond adequately to the mental health needs of seniors has been questioned and cost-effective solutions are required. Because the therapist's role in GSH is limited to supporting the patient, it is conceivable that this role could be assumed by trained and supervised lay providers (LP) instead of licensed providers. If this approach is effective, it could help provide many older adults with much needed mental health treatment at a lower cost. The main objective of this project is to evaluate the effectiveness of GSH guided by LP for GAD in older adults. Participants will be assigned randomly to an experimental group, which will receive treatment immediately, or to a control group whose treatment will be delayed. Data will be obtained through clinician evaluations and self-assessment questionnaires. They will include socio-demographic characteristics, symptoms of GAD, variables related to anxiety, such as depression and sleep difficulties, and participants' perception of treatment. For the experimental group, data collection will take place at four different times: before treatment begins, after treatment ends, and at 6 and 12 months after the end of treatment. Control group participants will be assessed on three occasions: before and after the waiting period and after receiving treatment. The efficacy of GSH will be established by comparing the change in the two groups on the main variables. We will also identify the characteristics of patients associated with improvement during treatment and document their perception of treatment.

DETAILED DESCRIPTION:
Few older adults with Generalized Anxiety Disorder (GAD) receive treatment although it is one of the most prevalent anxiety disorders in this population and involves significant health care costs. Studies show that older adults generally prefer psychotherapy and find it more acceptable than medication for help with anxiety. Unfortunately, face-to-face psychotherapy is difficult to access for many of them. Guided self-help (GSH) is an alternative to psychotherapy which requires that the patient take home a standardized psychological treatment and work through it more or less independently. The role of the therapist is primarily of supportive nature and the amount of contact between the patient and therapist is minimized. There is evidence that GSH based on the principles of cognitive-behavioral therapy (GSH-CBT) and guided by a licensed mental health provider is effective for treating GAD in older adults. However, the capacity of our health care system to respond adequately to the mental health needs of older adults has been questioned and cost-effective solutions are required to meet the needs of a rapidly aging population. Because the therapist's role in GSH-CBT is limited to supporting the patient, it is conceivable that this role could be assumed by trained and supervised lay providers (LP) instead of licensed providers. LP are generally providers with no post-graduate training in a specialized mental health program. The main goal of the study is to evaluate the efficacy of GSH-CBT guided by LP for GAD in older adults. Secondary goals are to identify the characteristics of patients associated with improvement during treatment and to document perception of treatment by patients and LP. We will conduct a multisite randomized controlled trial comparing an experimental group receiving GSH-CBT guided by LP to a wait-list control group. LP training will include readings, didactic training, and role plays. LP will be supervised throughout the project by licensed psychologists. Treatment will last 15 weeks and be based on a participant's manual. Weekly telephone sessions with LP (30 minutes maximum) will be limited to providing support. Data will be obtained through clinician evaluations and self-assessment questionnaires. They will include symptoms of GAD and variables related to anxiety, such as depression. For the experimental group, measurements will take place at pre- and post-treatment and at 6 and 12 months post-treatment. For the control group, three evaluations are planned: two pre-treatment evaluations (before and after the waiting period) and after receiving treatment (post-treatment). The efficacy of GSH-CBT will be established by comparing the change in the two groups on the main variables. This project will provide evidence on the effectiveness of a novel approach to treat GAD in older adults. If effective, it may be implemented on a larger scale and provide many older adults with much needed mental health treatment through an expanded workforce.

ELIGIBILITY:
Inclusion Criteria:

* 60 years of age or older
* meet at least criteria for subthreshold GAD at screening based on items of the Worry and Anxiety Questionnaire
* meet DSM-5 criteria for primary threshold or subthreshold GAD
* be able to read and speak French and to use the telephone without difficulty
* if an anxiety medication is used, commit to maintaining the type of medication or dose during eight weeks prior to treatment and during the protocol.

Exclusion Criteria:

* a disabling physical disorder that is not adequately controlled (e.g., acute heart disease, recent stroke)
* the presence of a substance use disorder
* presenting a bipolar disorder or symptoms of a psychotic disorder
* having significant cognitive impairment (score of less than 22 on the Telephone version of the Mini-Mental State Examination)
* currently receiving or having received psychotherapy for anxiety over the last six months.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Change in Penn State Worry Questionnaire | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  16 items rated on a scale ranging from 1 to 5. A higher total score indicates a greater tendency to worry.
Change in GAD-7 | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  7 items answered on a scale ranging from 0 to 3. A higher total score suggests greater severity.

SECONDARY OUTCOMES:
Change in Intolerance to Uncertainty Inventory | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  27 items rated on a scale ranging from 1 to 5. A higher total score suggests higher intolerance to uncertainty.
Change in Negative Problem Orientation Questionnaire | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  12 items rated on a scale ranging from 1 to 5. A higher total score suggests more negative attitudes toward problems.
Change in Cognitive Avoidance Questionnaire | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  25 items rated on a scale ranging from 1 to 5. A higher total score suggests more likely use of cognitive avoidance.
Change in Why Worry Questionnaire | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  25 items rated on a scale ranging from 1 to 5. A higher total score suggests a greater belief that worrying is useful.
Change in Geriatric Anxiety Inventory | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  20 items rated as "agree" or "disagree". Minimum score = 0; Maximum score = 20. A higher total score is indicative of greater severity of symptoms.
Change in Geriatric Depression Scale | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  30 items rated as "yes" or "no". Minimum score = 0; Maximum score = 30.A higher total score is indicative of greater severity of symptoms.
Change in Insomnia Severity Index | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  7 items rated on a scale ranging from 1 to 4. A higher total score suggests more severe insomnia.
Change in Sheehan Disability Scale | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  Three self-rated items of family, work, and social impairment rated on a scale ranging from 0 to 10.
Change in Mini-Mental State Examination, telephone version | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  Items on orientation to time and place, registration, attention, recall, and language. Scores vary between 0 and 26 with higher scores indicating better cognitive functioning.
Change in GAD diagnosis | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  The Anxiety and Related Disorders Interview Schedule for DSM-5 is a validated structured interview used to confirm the presence or absence of anxiety disorders and associated psychiatric diagnoses.

OTHER OUTCOMES:
Evaluation of treatment by participants | Post treatment (15 weeks)
  Measures participant's perception of treatment. 19 statements covering various aspects of treatment (modules, readings, exercises, telephone sessions, workload, organization and duration of treatment, and its usefulness). Each statement is evaluated on a four-point scale ranging from "strongly agree" to "absolutely disagree". A fifth possible answer, 'does not apply', is also provided.
Questionnaire of behavioral manifestations linked to anxiety | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  Twenty-four items evaluating six behaviors related to generalized anxiety, namely reassurance seeking, avoidance, control, procrastination, overplanning and checking. Items are rated on a five point Likert scale
Nine items relating to COVID-19 | Baseline, post treatment (15 weeks), 6 months and 12 months follow-up.
  These items were added to describe the reality of the participants while considering the effects of the pandemic on their anxiety. Five questions are framed as "yes or no" with an open-ended description of their answer choice whereas four items are rated on a five-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Centre de recherche de l'Institut universitaire de gériatrie de Montréal, Montreal, Quebec
  - École de psychologie, Université Laval, Québec, Quebec
  - Département de psychologie, Université de Sherbrooke, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Landreville P, Gosselin P, Grenier S, Carmichael PH. Self-help guided by trained lay providers for generalized anxiety disorder in older adults: study protocol for a randomized controlled trial. BMC Geriatr. 2021 May 22;21(1):324. doi: 10.1186/s12877-021-02221-x. PMID 34022795